CLINICAL TRIAL: NCT06564493
Title: A Prospective, Open-label, Randomized Controlled, Multicenter Clinical Study of Matched Sibling Donor Hematopoietic Stem Cell Transplantation Using a TBI or TMLI Conditioning Regimen for Pediatric Lymphoblastic Leukemia
Brief Title: A Prospective, Open-label, Randomized Controlled, Multicenter Clinical Study of MSD-HSCT Using a TBI or TMLI Conditioning Regimen for Pediatric ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xiangbo Wan, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-0213
Record Dates: First submitted 2024-07-04; First posted 2024-08-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMLI conditioning group (Experimental): Total Marrow, Central Nervous System and Lymphoid Irradiation (TMLI) plus Cyclophosphamide
  Interventions: Radiation: TMLI; Drug: Cyclophosphamide
- TBI conditioning group (Active Comparator): Total Body Irradiation (TBI) plus Cyclophosphamide
  Interventions: Radiation: TBI; Drug: Cyclophosphamide

INTERVENTIONS:
Radiation: TBI — The total dose of TBI is 12 Gy, administered on days -7, -6, and -5, with 2 Gy per fraction, twice daily, for a total of 6 fractions.
  Arms: TBI conditioning group
Radiation: TMLI — The total dose of TMLI is 12 Gy, administered on days -7, -6, and -5, with 2 Gy per fraction, twice daily, for a total of 6 fractions.
  Arms: TMLI conditioning group
Drug: Cyclophosphamide — The total dose of cyclophosphamide is 120 mg/kg, administered over 2 days on days -4 and -3.
  Other Names: CTX

SUMMARY:
This study aims to compare the effects of two different conditioning regimens on patients with acute lymphoblastic leukemia (ALL) undergoing matched sibling donor hematopoietic stem cell transplantation (MSD-HSCT): Total Body Irradiation (TBI) and Total Marrow, Central Nervous System and Lymphoid Irradiation (TMLI). Both regimens are supported and recommended by literature; however, there is no definitive evidence favoring one over the other. We hypothesize that the TMLI regimen, compared to the TBI regimen, may more effectively eliminate leukemia cells in the bone marrow and lymphoid tissues, thereby reducing the risk of relapse, while also minimizing damage to normal tissues, thus reducing conditioning-related toxicity and transplant-related mortality. This study aims to provide evidence for the optimal conditioning regimen for MSD-HSCT in pediatric ALL patients, with the goal of improving patient quality of life and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: Participants or guardians must voluntarily sign a written informed consent form.
2. Age and Gender: Participants should be male or female, aged 1-17 years, inclusive.
3. Diagnosis: Participants must be diagnosed with acute lymphoblastic leukemia (ALL) according to World Health Organization (WHO) criteria, and the diagnosis must apply to pediatrics aged 1-17 years.
4. Remission Status: The participant's leukemia must be in hematologic remission (complete remission, CR) prior to transplantation.
5. Donor Availability: There must be a suitable matched sibling donoravailable, and the participant must consent to undergo MSD hematopoietic stem cell transplantation (MSD-HSCT).
6. Karnofsky Performance Status: The participant must have a Karnofsky score of 70 or higher, indicating that they are capable of caring for themselves and carrying out normal activities. Additionally, they must not have significant organ dysfunction, defined by the following:

   * Cardiac Function: New York Heart Association (NYHA) classification of class II or lower.
   * Liver Function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels should be no more than 2.5 times the upper limit of normal. Bilirubin levels should be no more than 2 times the upper limit of normal.
   * Renal Function: Serum creatinine levels should be no more than 1.5 times the upper limit of normal, or the creatinine clearance rate should be at least 60 ml/min. o Pulmonary Function: Participants should not experience significant dyspnea, should not require oxygen therapy, should not have interstitial lung disease, and should not have any active pulmonary infections.

Exclusion Criteria: To be eligible for inclusion in the study, participants must not meet any of the following criteria:

1. The patient has not achieved hematologic remission before transplantation. 2. The patient has chosen a non-MSD donor.

3. The patient has severe cardiac, hepatic, renal, or pulmonary diseases that make them unable to tolerate the conditioning regimen.

4. The patient has an active or refractory infection, or other life-threatening complications.

5. The patient has a history of other malignant tumors, psychiatric disorders, or HIV infection.

6. The patients or guardians refuses to sign the informed consent form, is unwilling to comply with clinical follow-up required by the study, or does not consent to the use of their data to support future research, project presentations, and clinical practices.

7. The investigator deems the patient unsuitable for participation in the study for any other reason.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 2 years
  RFS is defined as the time from transplantation to the first relapse or death, with RFS is defined as the time from transplantation to the first relapse or death, with the date of the last follow-up as the endpoint.
acute Graft Versus Host Disease (aGVHD) | 100 days
  The incidence of aGVHD within 100 days post-transplant.
Overall Survival (OS) | 2 years
  OS is defined as the time from transplantation to death, with the date of the last follow-up as the endpoint.

SECONDARY OUTCOMES:
Transplantation Related Mortality (TRM) | 2 years
  The incidence of TRM in 2 years.
Relapse Rate (RR) | 2 years
  The incidence ratio of leukemia relapse in 2 years.
Conditioning-related Adverse Events (CRAE) | 30 days
  Based on CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No